CLINICAL TRIAL: NCT03410784
Title: A Phase II Clinical Trial of Pembrolizumab in Combination With Carboplatin-paclitaxel in Patients With Advanced (Stage III B-C-IV) Ovarian, Primary Peritoneal and Fallopian Tube Cancer: MITO28/MANGO OV4 Study
Brief Title: Pembrolizumab With Chemotherapy in Front Line Advanced Ovarian, Primary Peritoneal and Fallopian Tube Cancer
Acronym: MITO28MaNGOov4
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITO28 / MaNGO ov4; 2016-003926-18 (EudraCT Number)
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: PD-L1 Expression; prognostic factors; predictive factors; Patient reported outcomes
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-line chemotherapy with pembrolizumab (Other): * Pembrolizumab 200 mg i.v. on Day 1 every 3 weeks for up to 22 cycles
  * Paclitaxel 175 mg/m2 on Day 1 every 3 weeks for up to 6 cycles
  * Carboplatin (AUC 5) on Day 1 every 3 weeks for up to 6 cycles
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg i.v. on Day 1 every 3 weeks up to 22 cycles
Drug: Paclitaxel — Paclitaxel 175 mg/m2 i.v. on Day 1 every 3 weeks up to 6 cycles
Drug: Carboplatin — Carboplatin (AUC 5) i.v. on Day 1 every 3 weeks for up to 6 cycles

SUMMARY:
This study is designed to assess the therapeutic efficacy and toxicity of the combination chemotherapy Paclitaxel and Carboplatin with Pembrolizumab in patients with advanced ovarian cancer. The main objective is to test whether the therapeutic intervention benefits the patient evaluating the number of subjects who are progression-free after 18 months from the beginning of the first line treatment.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

* Have a histologically confirmed diagnosis of advanced (FIGO stage IIIB, IIIC, IV) epithelial ovarian, primary peritoneal or fallopian tube cancer.
* Have evidence of residual tumor after debulking surgery OR be non-eligible neither for primary surgery nor for neoadjuvant chemotherapy followed by interval debulking surgery
* Be willing and able to provide written informed consent/assent for the trial.
* Be at least 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Have tumor samples available for biomarker analysis.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Must be not eligible to receive Bevacizumab in combination with carboplatin and paclitaxel, due to contraindication, patient refusal or investigator choice
* Demonstrate adequate organ function

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent or investigational device and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to Pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (Grade 0 or 1 at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (Grade 0 or 1 at baseline) from adverse events due to a previously administered agent.

Note: Subjects with Grade 1 or 2 neuropathy are an exception to this criterion and may qualify for the study.

Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 28 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or other co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137) or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients free from progression | 18 months from beginning of first line treatment

SECONDARY OUTCOMES:
progression free survival | 3 years
overall survival | 5 years
number of patients with complete and partial responses | 18 months
worst grade toxicity per patient | evaluated every 3 weeks up to 18 months
  according to Common Toxicity Criteria for Adverse Events v. 4.03
changes in patient-reported outcome (PRO) scores of disease-related symptoms from baseline | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Nicoletta Colombo, M.D., Principal Investigator — European Institute of Oncology; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Gennaro Daniele, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (13):
- Italy (13):
  - Ospedale Generale Regionale "F. Miulli ", Acquaviva delle Fonti
  - Istituto Tumori Giovanni Paolo II, Bari
  - Spedali Civili - Università di Brescia, Brescia
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Nazionale Tumori, Milan
  - AOU Policlinico Federico II, Napoli
  - AOU Università degli studi della Campania "Luigi Vanvitelli", Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Ospedale Silvestrini, Perugia
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Universitario Gemelli Università Cattolica del Sacro Cuore, Roma